CLINICAL TRIAL: NCT06044688
Title: EyeQue VisionCheck 510(k) Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EyeQue Corp. (Industry)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EYEQUE-011
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Refractive Errors; Astigmatism
Keywords: Myopia; Hyperopia
MeSH Terms: conditions — Refractive Errors; Astigmatism; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Clinical site staff are masked to VisionCheck results. Participants are masked to VisionCheck and phoropter refraction measurements. The eyecare professionals performing Visit 2 refraction readings are masked to Visit 1 screening refraction readings.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Phoropter (Experimental): Refraction performed by an eye care professional using a phoropter.
  Interventions: Device: Phoropter
- VisionCheck (Active Comparator): Self-administered refraction performed using the EyeQue VisionCheck device.
  Interventions: Device: EyeQue VisionCheck

INTERVENTIONS:
Device: EyeQue VisionCheck — Automated subjective refraction system provides estimates of sphere, cylinder, and axis measurements of the eye.
  Arms: VisionCheck
Device: Phoropter — Standard of care, ophthalmic testing device, used by eye care professionals to measure the refractive error of the eye and determine prescription.
  Arms: Phoropter

SUMMARY:
Demonstrate that refraction measurements from the device agree with refraction measurements from a phoropter within clinically meaningful limits.

DETAILED DESCRIPTION:
The primary purpose of this study is to attain scientific objective evidence to support the VisionCheck Indications for Use by demonstrating that refraction measurements from the device agree with refraction measurements from a phoropter within clinically meaningful limits. The Indications for Use are:

"The EyeQue VisionCheck automated subjective refraction system provides an estimate of sphere, cylinder, and axis measurements of the eye"

Furthermore, the purpose of this study is to attain scientific objective evidence regarding the precision of the VisionCheck device.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet the following criteria to be enrolled in this study:

1. Participant or legally authorized representative (LAR) is willing and able to give informed consent
2. Participant is willing and able to follow all study procedures and requirements
3. Participant is able to use a smartphone
4. Participant is interested in getting refraction correction measurement
5. Participant is able to speak, read and write English fluently

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

1. Spherical correction >+8D or <-10D (outside the range of the VisionCheck measurement)
2. Astigmatism correction of less than -5D (optometric notation, outside the range of the VisionCheck measurement)
3. Inability to see the red and green lines (may be overlapped to form a, partially, yellow line) through the VisionCheck device
4. Participant does not have the physical dexterity to properly operate the EyeQue VisionCheck device or the EyeQue app on the smartphone in the Investigator's opinion
5. Has initiated any new medication in the two weeks prior to enrolling in this study that, in the best medical judgment of the Investigator, would impact their participation in the study or ability to use the EyeQue VisionCheck device
6. Eye surgery within 12 months prior to enrolling in this study (including Lasik or lens replacement)
7. Using anticholinergic medications (including first-generation antihistamines) or other medications known to affect vision within the greater of three days or five half-lives prior to enrolling in this study
8. Using an investigational drug or approved therapy for investigational use within the greater of three days or five half-lives prior to enrolling in this study
9. Color deficiency (Ishihara pseudoisochromatic plates: Concise 14-plate edition: six or more errors on plates 1-11; the 24-plate edition: seven or more errors on plates 1-15; the 38-plate edition: nine or more errors on plates 1-21)
10. Neurological and developmental conditions that may affect the outcome of the trial including, but not limited to, Multiple Sclerosis (MS), Stroke, Traumatic Brain Injury (TBI), Parkinson's Disease, Alzheimer's Disease, Dementia, Migraines, Optic Neuropathies, Brain Tumors, Hereditary Conditions (such as Leber's hereditary optic neuropathy (LHON) or retinitis pigmentosa), Epilepsy, Diplopia. Investigator discretion shall be applied to any additional conditions not listed.
11. Eye pathologies, including but not limited to:

    1. Glaucoma
    2. Any macular disease including macular degeneration, macular hole, macular dystrophy, epiretinal membrane, retinal vein occlusion, macular telangiectasia, central serous chorioretinopathy and cystoid macular edema
    3. Eye infection (corneal ulcer, corneal infiltrates, superficial punctate keratitis, ocular histoplasmosis syndrome)
    4. Keratoconus
    5. Diabetic neuropathy/retinopathy
    6. Cytomegalovirus retinitis
    7. Diabetic macular edema (evidence of fluid)
    8. Retinitis pigmentosa
    9. Amblyopia (best corrected visual acuity [BCVA] ≥ 20/30)
    10. Chronic or acute uveitis (cells and/or flare in the anterior chamber)
    11. Strabismus (manifest/latent, exotropia, esotropia, hypertropia, exophoria, and esophoria)
    12. Abnormal astigmatism (mild to severe, > 4D)
    13. Binocular vision anomalies
    14. Chronic dry eye
    15. Monovision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Assess agreement between the VisionCheck refraction measurement and a phoropter (standard of care) refraction measurement. | 3 months
  Bland-Altman limits of agreement (LoA) for within-eye differences between refraction measurements of sphere, cylinder, and axis obtained from VisionCheck and the subjective phoropter
Assess total variability and variance components for between- replicates (repeatability) and between-device/operator while adjusting for between-participant and between-site variability. | 3 months
  Percent coefficient of variation (%CV) and standard deviation (SD) of refraction measurement outputs in the form of sphere, cylinder, and axis obtained from VisionCheck

SECONDARY OUTCOMES:
Assess improvement in visual acuity brought forth by the VisionCheck refraction measurement. | 3 months
  95% upper prediction limit of improvement in visual acuity from refraction measurements obtained from VisionCheck compared to best corrected visual acuity from the subjective phoropter
Assess the safety of the VisionCheck device. | 3 months
  Adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), serious adverse device effects (SADEs), anticipated and unanticipated serious adverse device effects (ASADEs and USADEs, respectively)

IPD SHARING:
Plan to Share IPD: No